CLINICAL TRIAL: NCT01067105
Title: A 6-Month Open-Label, Long-Term Safety Extension Study of Once Daily Ciclesonide HFA Nasal Aerosol (160 μg) in The Treatment of Perennial Allergic Rhinitis (PAR) in Subjects 12 Years and Older
Brief Title: A 6 Month Study of Once Daily Ciclesonide Hydrofluoroalkane (HFA) Nasal Aerosol in The Treatment of Perennial Allergic Rhinitis (PAR) in Subjects 12 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060-635
Record Dates: First submitted 2010-02-09; First posted 2010-02-11 (Estimated); Results first posted 2012-06-11 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Perennial Allergic Rhinitis
Keywords: Perennial allergic rhinitis; allergic rhinitis; ciclesonide
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ciclesonide (Experimental): ciclesonide HFA 160 μg once daily
  Interventions: Drug: ciclesonide HFA 160 μg

INTERVENTIONS:
Drug: ciclesonide HFA 160 μg — ciclesonide HFA 160 μg once daily

SUMMARY:
6-month safety extension study in subjects who have completed Study 060-633 (NCT00953147). Evaluating the long-term safety of ciclesonide HFA nasal aerosol 160 μg administered once-daily in patients with Perennial Allergic Rhinitis.

DETAILED DESCRIPTION:
This is a 6-month multi-center, open-label, long-term safety extension study in subjects who have completed Study 060-633 (NCT00953147). This study is designed to evaluate the long-term safety of ciclesonide HFA nasal aerosol 160 μg administered once-daily to male and female subjects 12 years or older diagnosed with perennial allergic rhinitis (PAR). This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Subject has successfully completed all visits of Study 060-633.
* Subject has given written informed consent and assent, including privacy authorization as well as adherence to concomitant medication withholding periods, prior to participation.
* Subject is male or female 12 years and older.
* Subject must be in general good health (defined as the absence of any clinically relevant abnormalities as determined by the Investigator) based on screening physical examination, clinical laboratory tests, and medical history.
* Subject, if female 65 years of age or younger, must have a negative urine pregnancy test (performed at Visit 1). Females of childbearing potential must be instructed to and agree to avoid pregnancy during the study and must use an acceptable method of birth control:

  1. An oral contraceptive, an intrauterine device (IUD), implantable contraceptive, transdermal or injectable contraceptive for at least 1 month prior to entering the study with continued use throughout the study and for thirty days following study participation.
  2. Barrier method of contraception, eg, condom and/or diaphragm with spermicide while participating in the study.
  3. Abstinence.

Exclusion Criteria:

* Female subject who is pregnant or lactating.
* History of physical findings of nasal pathology, including nasal polyps.
* Subject has any condition that, in the judgment of the investigator, would preclude the subject from completing the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 824 (Actual)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (43):
  - Allergy and Asthma Specialists Group, Huntington Beach, California
  - California Allergy and Asthma Medical Group, Los Angeles, California
  - Southern California Research, Mission Viejo, California
  - CHOC PSF, AMC, Division of Allergy Asthma and Immunology, Orange, California
  - California Allergy and Asthma Medical Group, Palmdale, California
  - Allergy Associates Medical Group, San Diego, California
  - Bensch Research Associates, Stockton, California
  - Asthma and Allergy Associates, PC, Colorado Springs, Colorado
  - Storms Clinical Research Institute, Colorado Springs, Colorado
  - Colorado Allergy and Asthma Centers, Denver, Colorado
  - DataQuest Medical Research, Lawrenceville, Georgia
  - Allergy and Asthma Consultants, Lilburn, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Atlanta Allergy and Asthma Clinic, Woodstock, Georgia
  - Clinical Research Center of Indiana, Indianapolis, Indiana
  - GR, Bethesda, Maryland
  - Northeast Medical Research Associates, Inc., North Dartmouth, Massachusetts
  - Respiratory Medicine Research Institute of Michigan, Ypsilanti, Michigan
  - The Clinical Research Center, St Louis, Missouri
  - Clinical Research Group of Montana, Bozeman, Montana
  - Allergy and Asthma Center of NC, High Point, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Toledo Center for Clinical Research, Sylvania, Ohio
  - Allergy and Ashtma Research Group, Eugene, Oregon
  - Baker Allergy, Asthma, and Dermatology Research Center, Lake Oswego, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - Valley Clinical Research, Bethlehem, Pennsylvania
  - Asthma and Allergy Research, Upland, Pennsylvania
  - Asthma, Nasal Disease, and Allergy Research Center of New England, Providence, Rhode Island
  - National Allergy, Asthma, and Urticaria Centers, Charleston, South Carolina
  - ISIS Clinical Research, Austin, Texas
  - Sirius Clinical Research, Austin, Texas
  - TTS Research, Boerne, Texas
  - Pharmaceutical Research and Consulting, Dallas, Texas
  - North Texas Institute for Clinical Trials, Fort Worth, Texas
  - Allergy and Asthma Associates, Houston, Texas
  - Kerrville Research Associates, Kerrville, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Western Sky Medical Research, Paso, Texas
  - Biogenics Research Institute, San Antonio, Texas
  - Southwest Allergy and Asthma Center, San Antonio, Texas
  - Sylvana Research, San Antonio, Texas
  - ASTHMA Inc., Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ciclesonide
Started | 824
Completed | 683
Not Completed | 141
Not completed — Adverse Event | 14
Not completed — Protocol Violation | 48
Not completed — Withdrawal by Subject | 36
Not completed — Lost to Follow-up | 6
Not completed — Physician Decision | 6
Not completed — Other | 31

BASELINE CHARACTERISTICS:
Arm/Group | Ciclesonide
Number analyzed (Participants) | 824
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 64
  Between 18 and 65 years | 743
  >=65 years | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 38.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 529
  Male | 295
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 160
  Not Hispanic or Latino | 664
  Unknown or Not Reported | 0
Race/Ethnicity [Number; unit: participants]
  White/Caucasian | 690
  Black or African American | 104
  Asian | 15
  American Indian or Alaska Native | 1
  Native Hawaiian or Other Pacific Islander | 3
  Other | 7
  Multiple | 4
Baseline AM Reflective Total Nasal Symptom Score (rTNSS) [Mean (Standard Deviation); unit: units on a scale] — TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization.
  units on a scale | 5.66 (3.07)
Baseline AM Instantaneous Total Nasal Symptom Score (iTNSS) [Median (Standard Deviation); unit: units on a scale] — TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, iTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Instantaneous TNSS measures these symptoms over the previous 10 minute time interval. Baseline was the average of the AM and PM responses obtained during the run-in period up to 6 days prior to randomization.
  units on a scale | 5.12 (3.05)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Experiencing Adverse Events (AEs)
Time Frame: Weeks 1-26
Population: Intent to Treat Population
Measure: Number; unit: percentage of participants
Arm/Group | Ciclesonide
Number analyzed (Participants) | 824
percentage of participants | 51.5

2. Primary Outcome: Percentage of Subjects Experiencing Serious Adverse Events (SAEs)
Time Frame: Weeks 1-26
Population: Intent to Treat Population
Measure: Number; unit: percentage of participants
Arm/Group | Ciclesonide
Number analyzed (Participants) | 824
percentage of participants | 1.8

3. Primary Outcome: Percentage of Subjects Who Discontinue Due to AEs.
Time Frame: Weeks 1-26
Population: Intent to Treat Population
Measure: Number; unit: percentage of participants
Arm/Group | Ciclesonide
Number analyzed (Participants) | 824
percentage of participants | 1.7

4. Secondary Outcome: Percentage of Subjects Experiencing Local Nasal AEs
Description: Local Nasal adverse events are defined as adverse events occurring in the middle ear, nose, throat, and upper respiratory tract down to the larynx, anatomic regions.
Time Frame: Weeks 1-26
Population: Intent to Treat Population
Measure: Number; unit: percentage of participants
Arm/Group | Ciclesonide
Number analyzed (Participants) | 824
percentage of participants | 29.4

5. Secondary Outcome: Change From Baseline in Daily Subject-reported AM Reflective TNSS Averaged Over the 6-month Treatment Period.
Description: TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval. Difference was calculated as the 6-month treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Baseline and Weeks 1-26
Population: Intent to Treat Population. Subjects with missing date were not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ciclesonide
Number analyzed (Participants) | 823
units on a scale | -0.50 (1.46)

6. Secondary Outcome: Change From Baseline in Daily Subject-reported AM Instantaneous TNSS Averaged Over the 6-month Treatment Period.
Description: TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, iTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Instantaneous TNSS measures these symptoms over the previous 10 minute time interval. Difference was calculated as the six month treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Baseline and Weeks 1-26
Population: Intent to Treat Population. Subjects with missing date were not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ciclesonide
Number analyzed (Participants) | 823
units on a scale | -0.54 (1.37)

7. Secondary Outcome: Change From Baseline in Daily Subject-reported AM Reflective TNSS at Each Month Over the 6-month Treatment Period.
Description: TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval. Difference was calculated as the month treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Baseline and Months 1, 2, 3, 4, 5, and 6
Population: Intent to Treat Population. Subjects with missing date were not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ciclesonide
Number analyzed (Participants) | 823
units on a scale
  Month 1 (n=823) | -0.18 (1.26)
  Month 2 (n=806) | -0.48 (1.49)
  Month 3 (n=768) | -0.64 (1.57)
  Month 4 (n=743) | -0.69 (1.70)
  Month 5 (n=716) | -0.64 (1.77)
  Month 6 (n=697) | -0.54 (1.87)

8. Secondary Outcome: Change From Baseline in Daily Subject-reported AM Instantaneous TNSS at Each Month Over the 6-month Treatment Period.
Description: TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, iTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Instantaneous TNSS measures these symptoms over the previous 10 minute time interval. Difference was calculated as the month treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Baseline and Months 1, 2, 3, 4, 5, 6
Population: Intent to Treat Population. Subjects with missing date were not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ciclesonide
Number analyzed (Participants) | 823
units on a scale
  Month 1 (n=823) | -0.26 (1.16)
  Month 2 (n=806) | -0.55 (1.41)
  Month 3 (n=768) | -0.66 (1.47)
  Month 4 (n=743) | -0.70 (1.57)
  Month 5 (n=716) | -0.67 (1.68)
  Month 6 (n=697) | -0.57 (1.73)

9. Secondary Outcome: Ratio (Reported as Percentage) of Correct Advances of the Dose Indicator Out of Expected Advances
Description: Ratio of correct advance is defined as the (number of doses actuated/number of doses reported) * 100% and therefore reported as a percentage.
Time Frame: Weeks 0-12
Population: Intent to Treat Population. Subjects with missing dosing indicator data were excluded from these analyses.
Measure: Mean (Standard Deviation); unit: percentage of correct advances
Arm/Group | Ciclesonide
Number analyzed (Participants) | 824
percentage of correct advances
  Week 0-6 (n=778) | 112.29 (23.64)
  Week 6-12 (n=732) | 112.23 (23.72)

10. Secondary Outcome: Number of Devices With Actuation Consistency
Description: Actuation consistency is defined as a dose indicator count within ±20% of the subject self report of study medication administration
Time Frame: Weeks 0-6 and 6-12
Population: Intent to Treat Population.
Measure: Number; unit: devices
Arm/Group | Ciclesonide
Number analyzed (Participants) | 824
devices
  Week 0-6 | 556
  Week 6-12 | 531

11. Secondary Outcome: Percentage of Devices With Actuation Consistency
Description: as for outcome 10
Time Frame: Weeks 0-6 and 6-12
Population: Intent to Treat Population
Measure: Number; unit: percentage of devices
Arm/Group | Ciclesonide
Number analyzed (Participants) | 824
percentage of devices
  Week 0-6 | 71.5
  Week 6-12 | 72.5

12. Secondary Outcome: Number of Devices With Major Discrepancies
Description: A major discrepancy is defined as a discrepancy of >20 actuations between the dose indicator and subject self report of study medication administration
Time Frame: Weeks 0-6 and 6-12
Population: Intent to Treat Population
Measure: Number; unit: devices
Arm/Group | Ciclesonide
Number analyzed (Participants) | 824
devices
  Week 0-6 | 144
  Week 6-12 | 117

13. Secondary Outcome: Percentage of Devices With Major Discrepancies
Description: as for outcome 12
Time Frame: Weeks 0-6 and 6-12
Population: Intent to Treat Population
Measure: Number; unit: percentage of devices
Arm/Group | Ciclesonide
Number analyzed (Participants) | 824
percentage of devices
  Week 0-6 | 18.5
  Week 6-12 | 16.0

14. Secondary Outcome: Number of Subjects Responding to the Subject Satisfaction Dose Indicator Survey
Description: Participants responding to a survey that consisted of 7 questions assessing subject satisfaction with the dose indicator.
Time Frame: Weeks 6 and 12
Population: Intent to Treat Population
Measure: Number; unit: participants
Arm/Group | Ciclesonide
Number analyzed (Participants) | 824
participants
  Week 6 | 794
  Week 12 | 744

ADVERSE EVENTS:
Arm/Group | Ciclesonide
Serious Adverse Events (participants affected / at risk) | 15/824
Other Adverse Events (participants affected / at risk) | 329/824
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciclesonide (N=824)
Artrial flutter (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Renal injury (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Troponin increased (Investigations) | 1 (1)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Mental status change (Psychiatric disorders) | 1 (1)
Endometrial hypertrophy (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Imprisonment (Social circumstances) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciclesonide (N=824)
Bronchitis (Infections and infestations) | 21 (24)
Nasopharyngitis (Infections and infestations) | 31 (35)
Sinusitis (Infections and infestations) | 38 (42)
Upper respiratory tract infection (Infections and infestations) | 61 (72)
Urinary tract infection (Immune system disorders) | 22 (23)
Viral upper respiratory tract infection (Infections and infestations) | 17 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (23)
Headache (Nervous system disorders) | 39 (56)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 46 (64)
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 13 (14)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 20 (21)

LIMITATIONS AND CAVEATS:
Open label study investigating a dose higher than the US FDA approved dose (74 mcg once daily) for allergic rhinitis subjects. Publication references to 148 mcg is equivalent to 160 mcg.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other